CLINICAL TRIAL: NCT04312997
Title: A Phase 2 Multiple Dose Study to Evaluate the Efficacy and Safety of PUL-042 Inhalation Solution in Reducing the Severity of COVID-19 in Adults Positive for SARS-CoV-2 Infection
Brief Title: The Use of PUL-042 Inhalation Solution to Reduce the Severity of COVID-19 in Adults Positive for SARS-CoV-2 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pulmotect, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PUL-042-502
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PUL-042 Inhalation Solution (Experimental): PUL-042 Inhalation Solution given by nebulization on Study Days 1, 3 and 6
  Interventions: Drug: PUL-042 Inhalation Solution
- Sterile saline for inhalation (Placebo Comparator): Sterile saline for Inhalation given by nebulization on Study Days 1, 3 and 6
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PUL-042 Inhalation Solution — 20.3 µg Pam2 : 29.8 µg ODN/mL (50 µg PUL-042)
  Arms: PUL-042 Inhalation Solution
Drug: Placebo — Sterile saline for inhalation
  Arms: Sterile saline for inhalation

SUMMARY:
Adults who have tested positive for SARS-CoV-2 infection and who may require supplemental oxygen will receive PUL-042 Inhalation Solution or placebo 3 times over a one week period in addition to their normal care. Subjects will be be followed and assessed for their clinical status over 28 days to see if PUL-042 Inhalation Solution improves the clinical outcome

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a positive test for SARS-CoV-2.
2. COVID-19 signs and symptoms such as (fever, cough, shortness of breath or fatigue) with onset within the 7 days prior to Screening
3. Subjects should be Ordinal Scale for Clinical Improvement score of 4 or less.
4. Subjects receiving oxygen should have pulse oximetry ≥ 93% on 3 liters per minute of oxygen or less delivered by nasal prongs.
5. Subjects can be receiving standard of care (SOC) for COVID-19, this includes marketed therapies or therapies with Emergency Use Authorization (EUA) for COVID-19 treatment.
6. Subject's spirometry (FEV1 and forced vital capacity [FVC]) must be ≥70% of predicted value.
7. If female, the subject must be surgically sterile or ≥ 1 year postmenopausal. If of child-bearing potential (including being < 1years postmenopausal) and, if participating in sexual activity that may lead to pregnancy, the subject agrees to use an effective dual method of birth control (acceptable methods include intrauterine device, spermicide, barrier, male partner surgical sterilization, and hormonal contraception) during the study and through 30 days after completion of the study.
8. If female, must not be pregnant, plan to become pregnant, or nurse a child during the study and through 30 days after completion of the study. A pregnancy test must be negative at the Screening Visit, prior to dosing on Day 1.
9. If male, must be surgically sterile or, if not surgically sterile and if participating in sexual activities that may lead to pregnancy, be willing to practice two effective methods of birth control (acceptable methods include barrier, spermicide, or female partner surgical sterilization) during the study and through 30 days after completion of the study.
10. Must have the ability to understand and give informed consent.

Exclusion Criteria:

1. No documented infection with SARS-CoV-2.
2. Patients who are in respiratory distress or require high flow oxygen, non-invasive ventilation or mechanical ventilation (Ordinal Scale for Clinical Improvement >4) or with pulse oximetry less than 93% on oxygen with a flow rate of 3 liters per minute or less by nasal prongs at the time of screening.
3. Known history of chronic pulmonary disease (e.g., asthma [including atopic asthma, exercise-induced asthma, or asthma triggered by respiratory infection], chronic pulmonary disease, pulmonary fibrosis, COPD), pulmonary hypertension, or heart failure.
4. Exposure to any investigational therapy (defined as any agent not currently marketed or without EUA) at the time of or within 30 days prior to the Screening Visit.
5. Any condition which, in the opinion of the Principal Investigator, would prevent full participation in this trial or would interfere with the evaluation of trial endpoints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Broom, MD, Study Director — Pulmotect, Inc.
Locations (11):
- United States (11):
  - University of California Irvine, Orange, California
  - Premeir Urgent Care of California, San Bernardino, California
  - Clinical Research of South Florida Alliance for Multispecialty Research, Coral Gables, Florida
  - Invesclinic US LLC, Fort Lauderdale, Florida
  - DBC Research Corp., Tamarac, Florida
  - Affinity Clinical Research, LLC, Tampa, Florida
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - Ascension St. John, Bartlesville, Oklahoma
  - Ascension St. John, Tulsa, Oklahoma
  - MD Anderson Cancer Center, Houston, Texas
  - Next Level Urgent Care, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PUL-042 Inhalation Solution | Sterile Saline for Inhalation
Started | 51 | 50
Completed | 45 | 47
Not Completed | 6 | 3

BASELINE CHARACTERISTICS:
Population: The number of Baseline Participants (99) differs from the numbers in the Participant Flow (101) as two participants were randomized but not treated. The ITT (Intent-to-treat) population is 99 total (49 for PUL-042, 50 for placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | PUL-042 Inhalation Solution | Sterile Saline for Inhalation | Total
Number analyzed (Participants) | 49 | 50 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 49 | 93
  >=65 years | 5 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (15.89) | 43 (11.86) | 42.6 (13.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 33 | 57
  Male | 25 | 17 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 30 | 59
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 3 | 5
  White | 45 | 42 | 87
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 49 | 50 | 99
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.55 (7.176) | 28.50 (7.594) | 28.52 (7.354)
Time from Symptom Onset to Day 1 Treatment [Mean (Standard Deviation); unit: days] | 6.3 (1.96) | 5.9 (1.92) | 6.1 (1.94)
FEV1 % Predicted [Mean (Full Range); unit: Percent] | 88.5 [72 to 111] | 94.2 [70 to 129] | 91.4 [70 to 129]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Worsening of COVID-19 Within 28 Days
Description: To determine the efficacy of PUL-042 Inhalation Solution in decreasing the severity of COVID-19 in subjects: 1) who have documented SARS-CoV-2 infection, and 2) if receiving oxygen, should have pulse oximetry ≥ 93% on 3 liters per minute of oxygen or less delivered by nasal prongs (Ordinal Scale for Clinical Improvement 4 or less) at the time of enrollment.
  The primary endpoint analysis is the evaluation of the number of patients with clinically meaningful worsening of COVID-19 within 28 days from the start of experimental therapy, as indicated by an increase of at least 2 points on the Ordinal Scale for Clinical Improvement (OSCI). The OSCI used in this study is derived from a draft scale proposed by the World Health Organization for clinical improvement. Higher values represent a worse outcome.
  The OSCI is a nine-point scale (0-8) with 0 being no clinical or virological evidence of infection and 8 being death.
Time Frame: 28 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PUL-042 Inhalation Solution | Sterile Saline for Inhalation
Number analyzed (Participants) | 49 | 50
Participants | 1 | 1

2. Secondary Outcome: Number of Participants With Positive SARS-CoV-2 Test Results at the End of Study
Description: SARS-Co-V-2 positivity up to 28 days from the start of experimental therapy.
Time Frame: 28 days
Population: Analysis Population: number of ITT (Intent-to-Treat) participants with non-missing test results (Positive or Negative) at the end of the study or early termination visit
Measure: Count of Participants; unit: Participants
Arm/Group | PUL-042 Inhalation Solution | Sterile Saline for Inhalation
Number analyzed (Participants) | 41 | 45
Participants | 8 | 9

3. Secondary Outcome: Number of Participants With Worsening of COVID-19 Over 14 Days
Description: To determine the difference in the proportion of COVID-19 patients with clinically meaningful worsening of COVID-19 within 14 days from the start of experimental therapy, as indicated by an increase of at least 2 points on the Ordinal Scale for Clinical Improvement (OSCI).
  The OSCI is a nine-point scale (0-8) with 0 being no clinical or virological evidence of infection and 8 being death.
Time Frame: 14 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PUL-042 Inhalation Solution | Sterile Saline for Inhalation
Number analyzed (Participants) | 49 | 50
Participants | 1 | 1

4. Secondary Outcome: Time to COVID-19 Symptom Improvement: Respiratory Symptoms
Description: To assess the progression of COVID-19 severity during the study as measured by the SARS-CoV-2 Symptom Score.
  The SARS-CoV-2 Symptom Score measures 3 elements on a 0-3 scale (cough, shortness of breath or difficulty breathing, and muscle aches or fatigue) ranging from 0 for none to 3 for severe. The fourth element is fever and it is rated on a 0-4 scale with 0 being no fever and 4 being life-threatening.
  The time to respiratory symptom improvement is measured in days. Time to improvement of symptoms was prospectively defined as the time from an initial symptom score of ≥1 to a reduction of ≥1 point. The time to improvement of symptoms was evaluated for each individual symptom listed above.
Time Frame: 28 days
Population: Analyzed was the number of ITT participants (total 99) with at least 1 symptom score of >=1 for one symptom (total 92).
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | PUL-042 Inhalation Solution | Sterile Saline for Inhalation
Number analyzed (Participants) | 45 | 47
Days | 6 [4 to 7] | 9 [5 to 11]

5. Secondary Outcome: Time to Resolution of COVID-19 Symptoms
Description: The time to resolution of COVID-19 symptoms during the study was measured by the SARS-CoV-2 Symptom Score: The SARS-CoV-2 Symptom Score measures 3 elements on a 0-3 scale (cough, shortness of breath or difficulty breathing, and muscle aches or fatigue) ranging from 0 for none to 3 for severe. The fourth element is fever and it is rated on a 0-4 scale with 0 being no fever and 4 being life-threatening.
  The time to the first occurrence of resolution of symptoms (in days) was defined as the time from the first symptom score of ≥1 to a symptom score of 0.
Time Frame: 28 days
Population: Analyzed was the number of ITT participants (total 99) with at least 1 symptom score of >=1 for one symptom (total 92).
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | PUL-042 Inhalation Solution | Sterile Saline for Inhalation
Number analyzed (Participants) | 45 | 47
Days | 11 [6 to 15] | 11 [9 to 15]

6. Secondary Outcome: Number of Participants Requiring ICU Admission
Description: The requirement for ICU admission within 28 days from the start of the experimental therapy.
Time Frame: 28 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PUL-042 Inhalation Solution | Sterile Saline for Inhalation
Number analyzed (Participants) | 49 | 50
Participants | 0 | 2

7. Secondary Outcome: Number of Participants Requiring Mechanical Ventilation
Description: The requirement for mechanical ventilation within 28 days from the start of the experimental therapy.
Time Frame: 28 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PUL-042 Inhalation Solution | Sterile Saline for Inhalation
Number analyzed (Participants) | 49 | 50
Participants | 0 | 0

8. Secondary Outcome: Number of Participant Death
Description: All-cause mortality at 28 days from the start of experimental therapy.
Time Frame: 28 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PUL-042 Inhalation Solution | Sterile Saline for Inhalation
Number analyzed (Participants) | 49 | 50
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Subjects will participate for 28 days.
Description: Reporting is done by organ system, irrespective of causality. The Safety Population Set (99) was defined as all randomized participants (101) who received at least one dose of experimental treatment (99) - PUL-042 (49) or Placebo (50), but participants were categorized based on the treatment actually received rather than as randomized. One subject was randomized to PUL-042 but incorrectly received Placebo, resulting in 48 participants receiving PUL-042 and 51 participants receiving Placebo.
Arm/Group | PUL-042 Inhalation Solution | Sterile Saline for Inhalation
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/51
Serious Adverse Events (participants affected / at risk) | 1/48 | 2/51
Other Adverse Events (participants affected / at risk) | 7/48 | 0/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PUL-042 Inhalation Solution (N=48) | Sterile Saline for Inhalation (N=51)
COVID-19 (Infections and infestations) | 1 | 2 — COVID-19 worsening
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PUL-042 Inhalation Solution (N=48) | Sterile Saline for Inhalation (N=51)
Nausea (Gastrointestinal disorders) | 3 | 0
Chest discomfort (General disorders) | 2 | 0
Chills (General disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/97/NCT04312997/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/97/NCT04312997/SAP_001.pdf